CLINICAL TRIAL: NCT05881408
Title: A Phase 3, Multinational, Randomized, Double-Blind, Placebo-Controlled Systemic Gene Transfer Therapy Study to Evaluate the Safety and Efficacy of SRP- 9001 in Non-Ambulatory and Ambulatory Subjects With Duchenne Muscular Dystrophy (ENVISION)
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety and Efficacy of Delandistrogene Moxeparvovec (SRP-9001) in Non-Ambulatory and Ambulatory Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: ENVISION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRP-9001-303; 2020-002372-13 (EudraCT Number); 2024-512626-28-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Gene-Delivery; Pediatric; North Star Ambulatory Assessment (NSAA); Performance of Upper Limb (PUL); Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delandistrogene Moxeparvovec followed by Placebo (Experimental): Participants will receive single IV infusion of delandistrogene moxeparvovec on Day 1. Then, participants will receive a single IV infusion of matching placebo at approximately 72 weeks.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo
- Placebo followed by Delandistrogene Moxeparvovec (Placebo Comparator): Participants will receive matching placebo IV infusion on Day 1. Then, participants will have the opportunity to receive a single IV infusion of delandistrogene moxeparvovec at approximately 72 weeks.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
Genetic: placebo — Single IV infusion of matching placebo

SUMMARY:
The study will evaluate the safety and efficacy of delandistrogene moxeparvovec gene transfer therapy in non-ambulatory and ambulatory males with DMD. This is a randomized, double-blind, placebo-controlled 2-part study. Participants will be in the study for approximately 128 weeks. All participants will have the opportunity to receive intravenous (IV) delandistrogene moxeparvovec in either Part 1 or Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of DMD based on documented clinical findings and prior genetic testing.
* Cohort 1 only: Non-ambulatory per protocol-specified criteria.
* Cohort 2 only: Ambulatory per protocol-specified criteria and ≥8 to <18 years of age at the time of Screening.
* Ability to cooperate with motor assessment testing.
* Stable daily dose of oral corticosteroids for at least 12 weeks prior to Screening, and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight).
* Recombinant Adeno-Associated Virus Serotype rh74 (rAAVrh74) antibody titers are not elevated as per protocol-specified requirements.
* A pathogenic frameshift mutation or premature stop codon in the DMD gene, except for any deletion mutations in exon 8 and/or 9.

Exclusion Criteria:

* Exposure to gene therapy, investigational medication, or any treatment designed to increase dystrophin expression within protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.
* Presence of any other clinically significant illness, medical condition, or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risk for gene transfer.

Other inclusion or exclusion criteria could apply.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change From Baseline in the Total Score of Performance of Upper Limb (PUL) (Version 2.0) at Week 72 | Baseline, Week 72

SECONDARY OUTCOMES:
Part 1: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 72 | Baseline, Week 72
Part 1: Change From Baseline in Percent Predicted Peak Expiratory Flow (PEF) at Week 72 | Baseline, Week 72
Part 1: Quantity of Delandistrogene Moxeparvovec Dystrophin Expression at Week 12 as Measured by Western Blot | Week 12
Part 1: Change From Baseline in Patient-Reported Outcomes Measurement Information (PROMIS) Score in Upper Extremity Function to Week 72 | Baseline, Week 72
Number of Participants with a Treatment Emergent Adverse Event (TEAE), Adverse Event of Special Interest (AESI), and Serious Adverse Event (SAE) | Baseline up to Week 124
Part 1 (For Cohort 2 Only): Change From Baseline in the North Star Ambulatory Assessment (NSAA) Total Score at Week 72 | Baseline, Week 72
Part 1: Change From Baseline in Global Circumferential Strain as Measured by Cardiac MRI at Week 72 | Baseline, Week 72
Part 1: Change From Baseline in the Middle Domain Score of PUL (Version 2.0) at Week 72 | Baseline, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (46):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - University of California at Davis Medical Center, Sacramento, California
  - Rady Children's Hospital-San Diego, San Diego, California
  - University of Florida, UF Health Center for Pediatric Neuromuscular and Rare Diseases, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Charlotte R. Bloomberg Children's Center, Pediatric Clinical Research Unit, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University of St. Louis, St. Louis Children's Hospital, St Louis, Missouri
  - University of Rochester, Department of Neurology, Rochester, New York
  - Lenox Baker Children's Hospital (Duke University), Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium
- Canada (3):
  - The Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Research Institute McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec - Université Laval (pavillon Centre Hospitalier Universitaire Laval), Québec
- Germany (3):
  - LMU- Klinikum der Universitat Munchen, Kinderklinik und Kinderpoliklinik im Dr. von Haunerschen Kinderspital, Abeteilung Neuropadiatrie, Campus Innenstadt, München, Bavaria
  - Universitatsklinikum Essen, Klinik fur Kinderheilkunde I, Abteilung Neuropadiatrie Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
- Hong Kong Children's Hospital, Hong Kong, Hong Kong
- Israel (2):
  - Institute of Neruology, Schneider Children's Medical Center of Israel, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - U.O.S.D Centro Traslazionale di Miologia e Patologie Neurodegenerative, Istituto G. Gaslini, Istituto Pediatrico di Ricovero e Cura a Carattere Scientifico, Genova
  - UOC Neurologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Neurologico Carlo Besta Neurepsichiatria Infantile 2 - Epilettologia e Neurologia dello Sviluppo, Milan
  - UOC Neuropsichiatria Infantile, Area Salute del Bambino, Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (3):
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi, Osaka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
- South Korea (4):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul, NAP
  - Kyungpook National University Hospital, Daegu
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Politecnic La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset/Astrid Lindgrens Barnsjukhus, Barnneurologen, Solna
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - Great Ormond Street Hospital for Children Foundation Trust, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Institute of Translational and Clinical Research, Newcastle upon Tyne

REFERENCES:
- See also: Click here to access the website, clinicaltrials.sarepta.com/ENVISION, for additional information for the study. — https://clinicaltrials.sarepta.com/ENVISION